CLINICAL TRIAL: NCT03615352
Title: Impact of Laparoscopic Ovarian Cystectomy Versus Aspiration and Coagulation on Ovarian Reserve and Pelvic Pain in Cases of Ovarian Endometrioma
Brief Title: Laparoscopic Ovarian Cystectomy Versus Aspiration and Coagulation in Ovarian Endometrioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaimaa Mostafa Mohammed Refaay El shemy (Other)
Responsible Party: Sponsor-Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Assistant lecturer of Obstetrics and Gynecology, Kasr Al ainy Hospital, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Laparoscopy in endometrioma
Record Dates: First submitted 2018-07-21; First posted 2018-08-03 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Endometrioma
Keywords: Endometrioma; laparoscopy; ovarian reserve; pelvic pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ovarian cystectomy (Experimental): laparoscopic ovarian cystectomy in endometrioma
  Interventions: Procedure: ovarian cystectomy
- ovarian cyst aspiration and coagulation (Experimental): laparoscopic ovarian endometrioma aspiration and coagulation
  Interventions: Procedure: ovarian cyst aspiration and coagulation

INTERVENTIONS:
Procedure: ovarian cystectomy — laparoscopic ovarian cystectomy in endometrioma
  Arms: ovarian cystectomy
Procedure: ovarian cyst aspiration and coagulation — laparoscopic ovarian cyst aspiration and coagulation in endometrioma
  Arms: ovarian cyst aspiration and coagulation

SUMMARY:
The aim of this study is to evaluate the impact of laparoscopic ovarian cystectomy versus aspiration and coagulation on ovarian reserve and pelvic pain in cases of ovarian endometrioma.

DETAILED DESCRIPTION:
All patients are presenting with ovarian endometrioma. They are all subjected to informed written consent, full history, general examination, local examination and transvaginal ultrasound. Follicular stimulating hormone (FSH), Lutenizing hormone (LH), Anti Mullerian hormone (AMH), Antral follicular count (AFC) and chronic pelvic pain which is assessed by Visual Analogue Scale (VAS) of pain scoring system ,all are to be determined before and after laparoscopic surgery (postoperative three months); for two groups (Group A) cystectomy and (Group B) aspiration and coagulation. Histopathological examination was done to the cystectomy group to confirm endometriosis and detect the presence of healthy ovarian tissue in the excised cyst wall.

ELIGIBILITY:
Inclusion Criteria:

* Female with age group 20-40 years.
* Female diagnosed by ultrasound with unilateral ovarian endometrioma ≥3cm.

Exclusion Criteria:

* Previous ovarian surgery.
* Endocrinological diseases affecting ovarian reserve e.g. Diabetes mellitus, hypothyroidism.
* Polycystic ovary syndrome (PCO).
* Suspicion of ovarian malignancy by ultrasound.
* Other pelvic pathology e.g. uterine fibroid, pelvic inflammatory disease (PID).
* High basal FSH >10mIU/mL (milli-international unit per milliliter).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Exploration of the impact of laparoscopic ovarian cystectomy versus aspiration and coagulation on Anti Mullerian hormone (AMH) as a measurement of ovarian reserve . | 3 months after laparoscopy
  Evaluation of ovarian reserve which is measured by Anti Mullerian hormone (AMH) in nano-gram per milliliter (ng/ml) before laparoscopy and after the surgery by 3 months.

SECONDARY OUTCOMES:
Exploration of the impact of laparoscopic ovarian cystectomy versus aspiration and coagulation on Antral Follicular Count (AFC) as a measurement of ovarian reserve. | 3 months after laparoscopy
  Evaluation of ovarian reserve by assessment of Antral Follicular Count (AFC) by measuring the number of visible ovarian follicles (2-10 mm mean diameter) that are observed during transvaginal ultrasonography in the early follicular phase (cycle days 2-5) in both ovaries. It is done before laparoscopy and after the surgery by 3 months.
Exploration of the impact of laparoscopic ovarian cystectomy versus aspiration and coagulation on chronic pelvic pain. | 3 months after laparoscopy
  Pelvic pain is measured by Visual analogue scale of pain (VAS) which is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10-cm scale).
  The pelvic pain is assessed before laparoscopy and after laparoscopy by 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Zayed Abd Elaziz, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt